CLINICAL TRIAL: NCT04606511
Title: Screening for Lymphedema
Brief Title: Lymphedema Screening
Acronym: LymphScreen
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Mads Gustaf Jørgensen, Principal Investigator, Odense University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: S-20200094
Record Dates: First submitted 2020-10-08; First posted 2020-10-28 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breast cancer patients with lymphedema (Other)
  Interventions: Diagnostic Test: Circumference tape measurements; Diagnostic Test: Indocyanine green lymphangiography; Diagnostic Test: bioimpedance spectroscopy; Diagnostic Test: Symptom score
- Breast cancer patients without lymphedema (Other)
  Interventions: Diagnostic Test: Circumference tape measurements; Diagnostic Test: Indocyanine green lymphangiography; Diagnostic Test: bioimpedance spectroscopy; Diagnostic Test: Symptom score

INTERVENTIONS:
Diagnostic Test: Circumference tape measurements — centimeter and volume criterias
Diagnostic Test: Indocyanine green lymphangiography — Presence of dermal backflow
Diagnostic Test: bioimpedance spectroscopy — 7.5 and 10 L-DEX criterias
Diagnostic Test: Symptom score — using lymph-icf, DASH and SF-36 questionnaires

SUMMARY:
Breast cancer-related lymphedema is one of the most common and feared consequences of breast cancer treatment. Currently, there is no established screening program for lymphedema. This cross-sectional study will investigate diagnostic modalities in screening for lymphedema in patients with and without known lymphedema after breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Previous breast cancer treated with axillary lymph node dissection
* No recurrence
* Understand the study
* Can talk, read and understand Danish

Exclusion Criteria:

* Pregnant or breast feeding
* Lymph node dissection from other basins
* Psychiatric disorder
* Not possible to perform indocyanine green lymphangiography

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
sensitivity, specificy, NPV and PPV | through study completion, approximately 1 year
  diagnosotic statistics of lymphedema measurements

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Plastic and Reconstructive Surgery, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Analytic Code
Time Frame: 5 years after study completion
Access Criteria: Upon reasonable request